CLINICAL TRIAL: NCT06965634
Title: Investigation of the Effectiveness of Lung Ultrasonography in the Management of Intraoperative Fluid Therapy, Prospective Observational Study
Brief Title: Investigation of the Effectiveness of Lung Ultrasonography in Intraoperative Fluid Management
Status: Not yet recruiting | Type: Observational
Sponsor: Korgün Ökmen (Other Government)
Responsible Party: Sponsor-Investigator, Korgün Ökmen, Principal Investigator, Bursa Yuksek Ihtisas Training and Research Hospital
Organization: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Other Study IDs: BursaYIEAH-2021-6-10
Record Dates: First submitted 2025-04-25; First posted 2025-05-11 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Intraoperative Fluid Management

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Lung ultrasound — Lung ultrasonography ; lung ultrasonography will be applied in 4 quadrants according to the LUS protocol and LUS score will be created.
  Other Names: Lung ultrasound score

SUMMARY:
Adequate and balanced fluid resuscitation is one of the cornerstones of intraoperative patient management. Over-resuscitation leading to positive fluid balance is associated with increased postoperative mortality and morbidity.

Invasive and non-invasive technologies can be used for the adequacy of intraoperative fluid therapy.

Lung ultrasonography (LUS) is a safe and accurate bedside imaging method. LUS, which is frequently used in the diagnosis of postoperative hypoxemia, has also begun to be preferred for fluid management in intensive care units.

DETAILED DESCRIPTION:
In this study, we aimed to investigate the effectiveness of intraoperative LUS data in the control of fluid therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with surgery with laparotomy

Exclusion Criteria:

* Chronic obstructive pulmonary disease
* Passed lung operation
* Uncontrolled hypertension
* Acute or chronic kidney failure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will undergo open surgery in ASA I-III risk classes.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-05-20 (Estimated); Primary Completion 2026-05-20 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
LUS | peroperative
  Lung ultrasound score (LUS) Lung ultrasonography; Lung ultrasound score will be created by performing ultrasonography in 4 quadrants according to the previously defined protocol.
  0 points indicated the presence of only A lines, less than 2 B lines
  1. point indicated 1-2 B lines
  2. points indicated the presence of more than 3 well-spaced B lines;
  3. points indicated the presence of combined B lines

SECONDARY OUTCOMES:
PVI | peroperative
  Pulse variable index (PVI) will be measured by finger pulse oximetry with the MASİMO device.
CVP | peroperative
  Central venous pressure(CVP)
  Pressure values measured by a central venous catheter applied by jugular or subclavian route
postoperative pulmonary complication | postoperative 6th hour
  hypoxia (partial oxygen pressure below 95 on pulse oximetry and 10% decrease from the initial value) atelectasis
biochemical data 1 | postoperative 6th hour
  glomerular filtration rate (GFR) values normal results range from 90 to 120 mL/min/1.73 m2.
biochemical data 2 | postoperative 6th hour
  Blood urea nitrogen value mg/dl
biochemical data 3 | postoperative 6th hour
  Blood creatinine value mmol/dl
Mechanical ventilation data 1 | peroperative
  End-Tidal Carbon Dioxide Pressure mm/hg The partial pressure of CO2 detected at the end of exhalation is between 35 and 45 mm Hg or 4.0 to 5.7 kPa.
Mechanical ventilation data 2 | peroperative
  Peak inspiratory pressure Values Peak inspiratory pressure is the highest pressure applied to the lungs during inhalation and should be kept below 35 cmH2O.It is automatically measured by respirators.
Mechanical ventilation data 3 | peroperative
  Tidal Volume value Tidal volume is the volume of gas moving into and out of the lungs with each breath. Normal tidal volume is 6 to 8 mL/kg, regardless of age. It is automatically measured by respirators.